CLINICAL TRIAL: NCT00514150
Title: Comparing Sodium Bicarbonate Plus Isotonic Normal Saline Versus Isotonic Normal Saline Alone to Prevent Contrast-Induced Nephropathy in Patients Undergoing Coronary Angiography: A Randomized Controlled Trial
Brief Title: Effect of Sodium Bicarbonate Solution in Decreasing the Incidence of Contrast Induced Nephropathy (CIN)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Collaborators: Tehran Heart Center (Other)
Responsible Party: Ali Vasheghani Farahani, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 85-02-30-3595(1)
Record Dates: First submitted 2007-08-08; First posted 2007-08-09 (Estimated); Last update posted 2008-09-05 (Estimated); Status verified 2008-09

CONDITIONS: Contrast Induced Nephropathy
Keywords: angiography; complications; contrast media; kidney; prevention
MeSH Terms: interventions — Sodium Bicarbonate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): 1075 cc of 154 mEq/L solution of NaCl 0.9% , prepared by adding 75 cc of 154 mEq/L NaCl 0.9 % to 1000 cc of 154 mEq/L NaCl 0.9%
  Interventions: Drug: normal saline 0.9%
- 2 (Active Comparator): 1075 cc fluid made by adding 75 cc of sodium bicarbonate 8.4% to 1000 cc of 154 mEq/ L NaCl 0.9%.
  Interventions: Drug: Sodium Bicarbonate plus normal saline 0.9%

INTERVENTIONS:
Drug: Sodium Bicarbonate plus normal saline 0.9% — IV sodium bicarbonate 8.4% solved in 154 mEq/ L NaCl 0.9% (infused at the rate of 3 ml/kg/ hour one hour before the angiographic procedure, continuing at the rate of 1 ml/kg/ hour for 6 hours after the procedure. Maximum rate of fluid permitted is that for a body weight of 110 Kg.
  Arms: 2
Drug: normal saline 0.9% — IV 154 mEq/L solution of NaCl 0.9% (infused at the rate of 3 ml/kg/ hour one hour before the angiographic procedure, continuing at the rate of 1 ml/kg/ hour for 6 hours after the procedure. Maximum rate of fluid permitted is that for a body weight of 110 Kg.)
  Arms: 1

SUMMARY:
Radio Contrast Induced Nephropathy (RCIN) remains a well recognized complication in patients undergoing diagnostic or interventional procedures requiring radiographic contrast agents. Recent studies have shown benefit in administering Sodium Bicarbonate over normal saline( the uniformly accepted prophylaxy) in preventing RCIN.Therefore the aim of the study is to evaluate the efficacy of sodium bicarbonate solved in normal saline compared with infusion of normal saline in prevention of RCIN.

DETAILED DESCRIPTION:
Radio Contrast Induced Nephropathy (RCIN) remains a well recognized complication in patients undergoing diagnostic or interventional procedures requiring radiographic contrast agents and is the third leading cause of acquired acute renal failure in hospitalized patients. Strategies for the prevention of radiocontrast nephropathy have focused on countering vasoconstriction (pre-hydration, fenoldopam, and theophylline), enhancing flow through the nephron (diuretics), or protection against oxygen-free-radical injury (urinary alkalinization and N-acetylcysteine).

Among all prophylactic measures that have been proposed, adequate preprocedural and postprocedural hydration has demonstrated effectiveness in the prevention of radiocontrast nephropathy. Thus, it remains the most frequently applied measure in clinical practice.

A Recent study in May 2004 have shown benefit in administering Sodium Bicarbonate over normal saline as a prophylaxy.Since alkalizing renal tubular fluid with bicarbonate may reduce injury.

Comparisons: IV 154 mEq/L solution of NaCl 0.9% OR IV 154 mEq/ L sodium bicarbonate solved in 154 mEq/ L NaCl 0.9%. Each fluid is infused at the rate of 3 ml/kg/ hour one hour before the angiographic procedure, continuing at the rate of 1 ml/kg/ hour for 6 hours after the procedure. Maximum rate of fluid permitted is that for a body weight of 110 Kg.

ELIGIBILITY:
Inclusion Criteria:

* individuals aged 18 years or older with stable serum creatinine levels of at least 1.5 mg/dl , who were scheduled to undergo diagnostic or therapeutic coronary artery angiography during the next 24 hours of hospitalization and were available until 5 days after the procedure for serum creatinine measurements.

Exclusion Criteria:

* serum creatinine levels of more than 8 mg/dl
* previous history of dialysis
* eGFR < 20
* emergency catheterization
* recent exposure to radiographic contrast agents (within previous two days of the study)
* radiocontrast agent dosage needed more than 300 cc during the procedure
* allergy to radiocontrast agent
* pregnancy
* administration of dopamine, mannitol , fenoldopam or N-Acetyl Cystein during the intended time of study
* need for continuous hydration therapy (e.g. sepsis )
* history of Multiple myeloma , Pulmonary edema , Uncontrolled hypertension (treated systolic blood pressure more than 160 mmHg, or diastolic blood pressure more than 100mmHg.) ,Severe heart failure (EF < 30% or NYHA 3-4).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2007-08; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
development of contrast induced nephropathy defined as an absolute (> or = 0.5 mg/dl) or relative increase (> or = 25%) in serum creatinine at 48 hours after exposure to a contrast agent compared to baseline serum creatinine values. | at 48 hours

SECONDARY OUTCOMES:
development of contrast induced nephropathy defined as an absolute (> or = 0.5 mg/dl) or relative increase (> or = 25%) in serum creatinine at 5 days after exposure to a contrast agent compared to baseline serum creatinine values. | at day 5
Days in hospital within the month post contrast | whithin the month post contrast
Urine PH after initial bolus | whithin 6 hours after initial bolus
development of contrast induced nephropathy defined as at least 25% decrease in glomerular filtration rate (GFR) at 48 hours. | at 48 hours
development of contrast induced nephropathy defined as at least 25% decrease in glomerular filtration rate (GFR) at day 5. | at day 5

CONTACTS AND LOCATIONS:
Overall Officials: Ali Vasheghani-Farahani, M.D., Study Director — Tehran University of Medical Sciences, Tehran Heart Center; Ebrahim Kassaian, M.D., Principal Investigator — Tehran Heart Center; Akbar Fotuhi, M.D., Principal Investigator — Tehran Heart Center; Mohammad Reza Khatami, M.D., Principal Investigator — Tehran Heart Center; Mojtaba Salarifar, M.D., Principal Investigator — Tehran Heart Center; Ahmad Iaminisharif, M.D., Principal Investigator — Tehran Heart Center; Saeid Sadeghian, M.D., Principal Investigator — Tehran Heart Center; Gholamreza Davoodi, M.D., Principal Investigator — Tehran Heart Center; Alireza Amirzadegan, M.D., Principal Investigator — Tehran Heart Center; Sirus Darabian, M.D., Principal Investigator — Tehran Heart Center; Gelareh Sadigh, M.D., Principal Investigator — Tehran University of Medical Sciences; Amir Hossein Razavi, M.D., Principal Investigator — Tehran University of Medical Sciences; Mohammad Ali Mansournia, MD, Principal Investigator — Tehran University of Medical Sciences; Mohammad Ali Boroumand, MD, Principal Investigator — Tehran Heart Center; Farah Aiatollahzade Esfehani, BSc,RN, Principal Investigator — Tehran Heart Center
Locations (1):
- Tehran Heart Center, Tehran, Iran